CLINICAL TRIAL: NCT00192257
Title: A Prospective, Randomized, Open-Label, Controlled Trial to Compare the Safety, Tolerability and Efficacy of Influenza Virus Vaccine, Trivalent, Type A&B, Live, Cold-Adapted (CAIV-T) With Influenza Virus Vaccine, Trivalent, Inactivated (TIV) in Children With Asthma Aged 6 Years to 17 Years
Brief Title: Trial to Compare the Safety, Tolerability and Efficacy of Influenza Virus Vaccine, (CAIV-T) With Influenza Virus in Children With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D153-P515
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Biological: CAIV-T and TIV

SUMMARY:
- Trial to assess asthma exacerbation through to the end of the study; and to demonstrate that the efficacy over one season against culture-confirmed influenza-illness; and finally to assess the safety and tolerability of CAIV-T in children with asthma.

DETAILED DESCRIPTION:
- To assess asthma exacerbation, being defined as acute wheezing illness associated with hospitalization, unscheduled clinic visits, or new prescriptions from study vaccination through to the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* who are aged at least 6 years to 17 years of age at the time of enrollment;
* with a clinical diagnosis of asthma by one of the following criteria:
* An International Classification of Diseases, Ninth revision (ICD-9) code 493 AND ≥one prescription for asthma medication;
* OR ≥one prescription for an inhaled beta-agonist and ≥one prescription for cromolyn;
* OR ≥Five prescriptions for any asthma medication (adapted from Kramarz et al,2000 and Osborne et al., 1995)1,2;
* asthma medication* is being defined as:
* inhaled and oral β -agonists
* theophyllin
* inhaled, oral and injected steroids
* other unclassified asthma medication
* antibiotics used for treatment of respiratory illness associated with a wheezing episode;
* at least one asthma medication should have been administered in the last 12 months
* who, if female and is post-menarche, has provided a negative pregnancy test prior to the study vaccination;
* who have provided written informed consent (as appropriate and according to national guidelines) and whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained;
* who, along with their parent(s)/legal guardian(s), will be available for duration of the trial;
* who/whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* who/whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids of a dose equivalent to a total of 20 mg/day or greater of prednisolone or equivalent, for more than 14 days duration until 2 weeks after corticosteroids have been discontinued 25;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* who have an immunosuppressed or an immunocompromised individual living in the same household;
* who received any influenza vaccine in the 6 months prior to enrollment, or are anticipated to receive a non-study influenza vaccine after enrollment;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the CAIV-T or TIV;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results;

Note: Pregnancy in any person who has regular contact with the subject is not a contraindication to the enrollment or ongoing participation of the subject in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2229
Dates: Start 2002-10; Study Completion 2003-05

PRIMARY OUTCOMES:
To demostrate that the efficacy over one influenza season against culture-confirmed influenza illness caused by community-acquired subtypes antifenically similar to those contained in the vaccine

SECONDARY OUTCOMES:
To demonstrate that the efficacy over one season of a single dose of CAIV-T was not inferior to that of one dose of TIV against culture-confirmed influenza-illness of any subtype
To compare the efficacy over a defined surveillance period against asthma exacerbations, asthma medication, clinical visits, hospitalizations, days off school (pharma-ecomonic measures) associated with influenza-like illness

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, M.D., Study Director — MedImmune LLC
Locations (2):
- Belgium (2):
  - Berchem
  - Brussels